CLINICAL TRIAL: NCT00453440
Title: Prospective Epidemiological Study of the Prevalence of HLA-B*5701 in HIV-1 Infected UK Patients
Brief Title: Prospective Epidemiological Study Of The Prevalence Of HLA-B*5701
Status: Completed | Type: Observational
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: CNA109479
Record Dates: First submitted 2007-03-28; First posted 2007-03-29 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: HIV; HLA-B*5701; Abacavir hypersensitivity reaction; HIV Infection
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; HIV Infections | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Cheek swab & blood test — Cheek swab & blood test

SUMMARY:
This is a study to determine the prevalence of a genetic marker, HLA-B5701, in the UK population. HLA-B*5701 has been strongly associated with the risk of an allergic reaction to a HIV medicine, Abacavir. The allergic reaction is known as a hypersensitivity reaction.

The study is a prospective study inviting HIV-1 positive patients over the age of 18 years to participate. Each participant will complete one study visit. They will be asked for details of their background including their age, sex, ethnicity, country of origin and parental country of origin.

They will be asked to give two samples to test for the presence of the genetic marker HLA-B*5701. The two samples are:

* A cheek swab
* A blood sample

In selected centres patients may be asked to provide up to two additional blood samples. These samples will be used to help develop and validate new methods of determining HLA-B*5701 testing.

ELIGIBILITY:
Inclusion criteria:

* HIV-1 infected patients over 18 years of age
* Patient willing & able to understand and provide written informed consent

Exclusion criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1502 (Actual)
Dates: Start 2007-03-20 (Actual); Primary Completion 2007-08-10 (Actual); Study Completion 2007-08-10 (Actual)

PRIMARY OUTCOMES:
Prevalence of HLA-B*5701 in the UK population via central labs | 2 Hours
  The widespread of HLA-B*5701 applied in the selected area in each participant of the UK population was tested via central labs. The result is summarized here.

SECONDARY OUTCOMES:
Prevalence of HLA-B*5701 in major UK ethnotypes in the study population. | 2 Hours
Description of HLA-B*5701 in the UK population via local labs. | 2 Hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (4):
- United Kingdom (4):
  - GSK Investigational Site, Woolwich, London, London
  - GSK Investigational Site, Birmingham, Warwickshire
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, London

REFERENCES:
- [Derived] Orkin C, Sadiq ST, Rice L, Jackson F; UK EPI team. Prospective epidemiological study of the prevalence of human leukocyte antigen (HLA)-B*5701 in HIV-1-infected UK subjects. HIV Med. 2010 Mar;11(3):187-92. doi: 10.1111/j.1468-1293.2009.00762.x. Epub 2009 Sep 24. PMID 19780860